CLINICAL TRIAL: NCT04386707
Title: A Randomized, Double-blinded, Controlled Clinical Trial to Evaluate Lot Consistency, Immunogenicity and Safety of Sabin Inactivated Polio Vaccine (Vero Cell) in 2-month-old Infants
Brief Title: Lot-consistency Clinical Trial of Sabin Strain Inactivated Polio Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-sIPV-3002
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Vaccine-lot 1 (Experimental): sIPV manufactured by Sinovac Biotech Co., Ltd at commercial scale.
  Interventions: Biological: Three doses of experimental sIPV of lot 1 at the schedule of 2,3,4 months of age
- Experimental Vaccine-lot 2 (Experimental): sIPV manufactured by Sinovac Biotech Co., Ltd at commercial scale.
  Interventions: Biological: Three doses of experimental sIPV of lot 2 at the schedule of 2,3,4 months of age
- Experimental Vaccine-lot 3 (Experimental): sIPV manufactured by Sinovac Biotech Co., Ltd at commercial scale.
  Interventions: Biological: Three doses of experimental sIPV of lot 3 at the schedule of 2,3,4 months of age
- Control Vaccine (Active Comparator): Wild strain IPV (wIPV）manufactured by Sanofi Pasteur S.A.
  Interventions: Biological: Three doses control wIPV at the schedule of 2,3,4 months of age

INTERVENTIONS:
Biological: Three doses of experimental sIPV of lot 1 at the schedule of 2,3,4 months of age — Three doses of experimental sIPV of lot 1 at the schedule of 2,3,4 months of age
  Arms: Experimental Vaccine-lot 1
Biological: Three doses of experimental sIPV of lot 2 at the schedule of 2,3,4 months of age — Three doses of experimental sIPV of lot 2 at the schedule of 2,3,4 months of age
  Arms: Experimental Vaccine-lot 2
Biological: Three doses of experimental sIPV of lot 3 at the schedule of 2,3,4 months of age — Three doses of experimental sIPV of lot 3 at the schedule of 2,3,4 months of age
  Arms: Experimental Vaccine-lot 3
Biological: Three doses control wIPV at the schedule of 2,3,4 months of age — Three doses control wIPV at the schedule of 2,3,4 months of age
  Arms: Control Vaccine

SUMMARY:
The purpose of this study is to evaluate the lot consistency, immunogenicity and safety of three lots of Sabin strain inactivated polio vaccine (Vero Cell) (sIPV) manufactured at commercial scale by Sinovac Biotech Co., Ltd., and evaluate the non-inferiority of investigational vaccine against a post-market inactivated polio vaccine.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, and positive-controlled clinical trial. A total of 1300 infants aged 2 months will be enrolled and assigned to 4 groups in a ratio of 1:1:1:1 to receive vaccination of 3 lots of investigational sIPV and control IPV manufactured by Sanofi Pasteur S.A respectively. Each subjects should finish the three-doses primary vaccination at the schedule of 2,3,4 months of age. Thirty-days safety observation after each dose of vaccination will be carried out. Venous blood should be collected from all the subjects before and 30 days after the three-doses primary vaccination, for the neutralizing antibody assay, and further to evaluate the immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 60-89 days;
* legal identity;
* Informed consent form has been signed by guardians.

Exclusion Criteria:

* Vaccination history of polio vaccine;
* Allergy history, history of asthma, including allergy history to vaccine or vaccine components, serious adverse reactions to the vaccine, such as urticaria, dyspnea, angioneurotic edema or stomachache, etc.;
* Congenital malformation or developmental disorder, genetic defect, serious malnutrition, etc.;
* Autoimmune disease or immunodeficiency/immunosuppression;
* Serious nervous system disorders (epilepsy, convulsion or tic) or mental disorders;
* Abnormal coagulation functions (such as coagulation factor deficiency, blood coagulation disease and blood platelet disorders) or obvious bruise or blood coagulation disorders diagnosed by the doctors;
* Receipt of immunosuppressant therapy, cytotoxic drug therapy and inhaled corticosteroid therapy (excluding the corticosteroid aerosol therapy for allergic rhinitis and surface corticosteroid therapy for acute non-complicated dermatitis);
* Receipt of blood products prior to this study;
* Receipt of other study drugs within 30 days prior to this study;
* Receipt of live attenuated vaccines within 14 days prior to this study;
* Receipt of subunit or inactivated vaccines within 7 days prior to this study;
* Acute diseases or acute exacerbation of chronic diseases within recent 7 days;
* Axillary temperature >37.0℃;
* Any other factors which are unsuitable for participation in the clinical trial as judged by the investigator.

Ages: 60 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1300 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-Geometric mean titer of neutralizing antibody | The 30th day after the third dose vaccination
  Micro-neutralization method will be used in the neutralizing antibody assay
Immunogenicity index-Seroconversion rates of neutralizing antibody | The 30th day after the third dose vaccination
  Micro-neutralization method will be used in the neutralizing antibody assay; Seropositive rates will be calculated based on the internationally accepted threshold value of ≥1:8. Seroconversion (1:8) is defined as a change from seronegative (<1:8) to seropositive (≥1:8) or a 4-fold increase from baseline titers if seropositive.

SECONDARY OUTCOMES:
Immunogenicity index-Seropositive rate of neutralizing antibody | The 30th day after the third dose vaccination
  Micro-neutralization method will be used in the neutralizing antibody assay; Seropositive rates will be calculated based on the internationally accepted threshold value of ≥1:8.
Immunogenicity index-Geometric mean ratio of neutralizing antibody | The 30th day after the third dose vaccination
  Micro-neutralization method will be used in the neutralizing antibody assay; Geometric mean ratio of neutralizing antibody titer after vaccination divided by that before vaccination
Safety index-Incidence of solicited adverse events | Day 0-7 after each dose vaccination, day 0 refers to the day of vaccination
  Solicited adverse events refer to the adverse events occur within day 0-7 after each dose vaccination with the solicited symptoms including injection-site induration, redness, swelling, rashes, or pruritus, and fever, allergic reactions, abnormal activity level, loss of appetite, nausea, vomiting and diarrhea.
Safety index-Incidence of unsolicited adverse events | Day 0-30 after each dose vaccination, day 0 refers to the day of vaccination
  Unsolicited adverse events refer to the unsolicited symptoms occur within day 0-7, and any symptoms occur out of that period
Safety index-Incidence of serious adverse events (SAEs) | From the beginning of vaccination to 30 days after the third dose vaccination
  SAEs refers to the events occur in the process of clinical trial which may need hospitalization, prolongation of hospitalization time, disability, dysfunction, be life-threatening or death or lead to congenital malformation.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zheng, Master, Principal Investigator — Yunnan Provincial Center for Disease Control and Prevention
Locations (4):
- China (4):
  - Yanshan County Center for Disease Control and Prevention, Wenshan, Yunnan
  - Qiubei County Center for Disease Control and Prevention, Wenshan, Yunnan
  - Mile City Center for Disease Control and Prevention, Yisa, Yunnan
  - Gejiu County Center for Disease Control and Prevention, Yisa, Yunnan

IPD SHARING:
Plan to Share IPD: No